CLINICAL TRIAL: NCT03011645
Title: Gene-by-Stress Interactions in Intervention Studies Significance
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of participants
Sponsor: Duke University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: Pro00070047; 2P01HL036587-25 (NIH)
Record Dates: First submitted 2017-01-04; First posted 2017-01-05 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases | interventions — ziprasidone; lorcaserin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Ziprasidone (Active Comparator): Ziprasidone 60 mg tablet by mouth, once a day for one day.
  Interventions: Drug: Ziprasidone
- Lorcaserin (Active Comparator): Lorcaserin 20 mg tablet by mouth, once a day for one day.
  Interventions: Drug: Lorcaserin
- Placebo Oral Tablet (Placebo Comparator): Sugar pill (in place of ziprasidone and lorcaserin) by mouth, once a day for one day.
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Ziprasidone — Given by mouth, single dose of 60 mg.
  Other Names: Geodon
  Arms: Ziprasidone
Drug: Lorcaserin — Given by mouth, single dose of 20 mg.
  Other Names: Belviq
  Arms: Lorcaserin
Drug: Placebo Oral Tablet — Given by mouth, single dose.
  Arms: Placebo Oral Tablet

SUMMARY:
The purpose of this study is to identify gene variants that increase risk of cardiovascular disease (CVD) and type 2 diabetes, particularly genes related to stress factors.

DETAILED DESCRIPTION:
In Aim 3, 100 subjects who participated in previous studies will be recruited to test the ability of a 5HTR2C agonist (lorcaserin) to increase and antagonist (ziprasidone) to reduce cortisol response to mental and metabolic stress in men carrying the rs6318 C allele and women in the rs6318 CC genotype of 5HTR2C. Lorcaserin is serotonin receptor agonist indicated for use as a weight loss drug. Ziprasidone is an antipsychotic indicated for treatment of bipolar disorder. Subjects will be treated with a single dose of each drug, 1 to 2 weeks apart, followed by a mental stress test and an oral glucose tolerance test with multiple blood draws. Each subject will also receive a placebo drug during one of the study visits.

ELIGIBILITY:
Inclusion Criteria:

* Men and women who have been enrolled in the STRRIDE, ENHANCED, and/or REMIT studies age 18 years or greater.
* Ability and willingness to provide informed consent.
* Individuals with specific genotypes as determined from our previous work on their samples through Aim 1 of this project.

Exclusion Criteria:

* Women who are known to be pregnant, intend to become pregnant, or breast-feeding will be excluded. Women who are of child bearing potential (under age 55) will be informed that they will need to have their urine tested for pregnancy and that they should not participate in the research if they are not willing to have the Investigators provide them with information on positive pregnancy test results. Subjects will be informed that the pregnancy testing is not being performed for clinical purposes and that the testing is not a substitute for their regular medical care if they need to know whether or not they may be pregnant.
* History of Type II diabetes mellitus.
* History of prolonged QT interval.
* Participation in an investigational drug trial within the last 30 days.
* Already taking either ziprasidone or lorcaserin or any potential confounding medications, for example, other weight loss medications or psychotropic medications.
* Unwillingness to fast for at least 6 hours prior to the research study visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2018-05-24 (Actual); Primary Completion 2020-01-28 (Actual); Study Completion 2020-01-28 (Actual)

PRIMARY OUTCOMES:
Change in peak blood cortisol during the metabolic stress of an OGTT | Baseline to 3-hours post OGTT
Change in peak blood cortisol during the metabolic stress of a mental stress test | Baseline to 3-hours post mental stress test

SECONDARY OUTCOMES:
Area-Under-the-Curve Glucose | Baseline to 2-hours post OGTT
Matsuda Insulin Resistance Index | Baseline to 2-hours post OGTT

CONTACTS AND LOCATIONS:
Overall Officials: William E Kraus, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No